CLINICAL TRIAL: NCT02154269
Title: Prospective, Double-blind, Randomized, Placebo-controlled Phase II Clinical Trial for Evaluation of G-CSF in Patients With Chronic Chagas Cardiomyopathy
Brief Title: Evaluation of G-CSF (Colony Stimulating Factor) in Patients With Chronic Chagas Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, PhD, Hospital Sao Rafael
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCL07/12
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Chronic Chagasic Myocarditis
Keywords: Chagas disease; G-CSF; Cell therapy
MeSH Terms: conditions — Chagas Disease | interventions — Therapeutics; Granulocyte Colony-Stimulating Factor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental): Subjects will be randomly assigned to receive treatment with G-CSF (10mg/kg/day) for five days, during 4 cicles.
  Interventions: Drug: Treatment with G-CSF (Granulocyte colony stimulating factor)
- Saline (Placebo Comparator): Subjects will be randomly assigned to receive saline for five days, during 4 cicles.
  Interventions: Drug: Placebo saline

INTERVENTIONS:
Drug: Treatment with G-CSF (Granulocyte colony stimulating factor) — Subjects will be randomly assigned to receive treatment with G-CSF (10mg/kg/day) for five days, during 4 cicles.
  Other Names: G-CSF
  Arms: G-CSF
Drug: Placebo saline — Subjects will be randomly assigned to receive treatment saline for five days, during 4 cicles.
  Other Names: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the effectiveness of treatment with G-CSF in patients with chronic heart failure secondary to Chagas disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chagas' disease confirmed by two serological tests with different methodologies;
* Diagnosis of Chagas' cardiomyopathy in NYHA functional classes II, III and IV of heart failure;
* Availability and willingness to participate, given the schedule of the study;
* Agreement and signing the written form.

Exclusion Criteria:

* Acute systemic infections
* Solid neoplasms, myelodysplastic syndrome, acute or chronic myeloid leukemia, confirmed by imaging studies or past medical history;
* Valvulopathies with hemodynamic consequences;
* Autoimmune, pulmonary, or degenerative diseases, confirmed by imaging studies or past medical history;
* Severe renal, hepatic or thyroid dysfunction, confirmed by imaging studies or past medical history;
* Pregnancy (confirmed by examination of β HCG) or lactation;
* Known hypersensitivity to G-CSF or to other components of the formula and / or hypersensitivity to proteins derived from E. coli.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
NYHA (New York Heart Association) functional class improvement | 6, 9 and 12 months after the therapy with G-CSF
  All patients will undergo periodic clinical evaluations in order to identify improvement on NYHA classification for heart failure.

SECONDARY OUTCOMES:
Assessment of cardiovascular function measured by transthoracic echocardiography | 6 and 12 months after the therapy
  All patients will be submitted to echocardiography after 6 and 12 months to assess improvements on ventricular function.
Assessment of cardiovascular function measured by cardiac magnetic resonance imaging | 12 months after therapy
  All patients will be submitted to a second cardiac magnetic resonance, after 12 months, to assess improvements on left ventricular ejection fraction.
Evaluation of functional capacity assessed by treadmill test and by 6-minute walk test | 12 months after the therapy
  All patients will be submitted to a second treadmill test and 6-minute walk test after 12 months to assess improvement on functional capacity.
Evaluation of improvement of quality of life | 6 and 12 months after the therapy
  All patients will respond to Minnesota Questionnaire to have an evaluation of quality of life after 6 and 12 months.
Determination of tolerability | 1, 5, 13, 17, 25, 29, 37 and 41 days and 3, 6, 9 and 12 months after the therapy
  All patients will be submitted to complete blood counts in several time frames in order to evaluate tolerability to G-CSF injection.

CONTACTS AND LOCATIONS:
Overall Officials: Milena BP Soares, PhD, Principal Investigator — Hospital São Rafael; Ticiana F Larocca, MD, Msc, Study Director — Hospital São Rafael; Ricardo Ribeiro-dos-Santos, PhD, Study Chair — Hospital São Rafael; Bruno SF Souza, MD, Msc, Study Chair — Hospital São Rafael; Márcia MN Rabelo, MD, Msc, Study Chair — Hospital São Rafael; Luís Cláudio L Correia, MD, Msc, Study Chair — Hospital São Rafael; Carolina T Macedo, MD, Msc, Study Chair — Hospital São Rafael; Clarissa LM Souza, MD, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Macedo CT, Larocca TF, Noya-Rabelo M, Aras R Jr, Macedo CRB, Moreira MI, Caldas AC, Torreao JA, Monsao VMA, Souza CLM, Vasconcelos JF, Bezerra MR, Petri DP, Souza BSF, Pacheco AGF, Daher A, Ribeiro-Dos-Santos R, Soares MBP. Efficacy and Safety of Granulocyte-Colony Stimulating Factor Therapy in Chagas Cardiomyopathy: A Phase II Double-Blind, Randomized, Placebo-Controlled Clinical Trial. Front Cardiovasc Med. 2022 Jun 9;9:864837. doi: 10.3389/fcvm.2022.864837. eCollection 2022. PMID 35757326